CLINICAL TRIAL: NCT04480372
Title: Overcoming Resistance to Immunotherapy Combining Gemcitabine With Atezolizumab in Advanced NSCLC and Mesothelioma Progressing Under Immune-checkpoint Inhibitors or Gemcitabine. A Multicenter, Single-arm, Open Label Phase II Trial With Two Cohorts
Brief Title: SAKK 17/18 (ORIGIN) MPM & NSCLC >1st Line Gemci & Atezo Ph II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 17/18
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Malignant Pleural Mesothelioma; Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; malignant pleural mesothelioma; Immunotherapy; Gemcitabine; Atezolizumab; phase II trial
MeSH Terms: conditions — Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; atezolizumab

STUDY DESIGN:
Intervention Model Description: A multicenter, single-arm, open label phase II trial with two cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSCLC (cohort 1) and inoperable MPM (cohort 2) (Experimental): Cohort 1 consists of NSCLC patients. Cohort 2 consists of MPM patients.
  Patients will be treated with gemcitabine at the dose of 1000 mg/m2 i.v. on day 1 and day 8 of each cycle (every 3 weeks) and with atezolizumab at the dose of 1200 mg i.v. on day 1 of each cycle (every 3 weeks).
  The trial treatments will be continued for max. 2 years or until discontinuation criteria are met (see Ch. 9.3), whichever occurs first. The follow-up phase will last up to 5 years from treatment start.
  Interventions: Drug: Gemcitabine; Drug: Atezolizumab

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine is administered at the dose of 1000 mg/m2 intravenously (i.v.) on day 1 and day 8 of each cycle (every 3 weeks).
Drug: Atezolizumab — Atezolizumab is administered at the dose of 1200 mg i.v. on day 1 of each cycle (every 3 weeks).

SUMMARY:
A significant number of patients with malignant pleural mesothelioma (MPM) and non-small cell lung cancer (NSCLC) are not cured with available treatments and will eventually relapse. After relapse treatment options are limited. Preclinical in vitro studies have demonstrated a synergism of immunotherapy with PD(L)1-targeting monoclonal antibodies and gemcitabine and ongoing clinical studies showed encouraging results.

The main objective of this trial is to determine the efficacy of chemotherapy (gemcitabine) combined with immunotherapy (atezolizumab) in patients with progressive NSCLC and MPM.

The trial treatments will be continued for max. 2 years or until discontinuation criteria are met. The follow-up phase will last up to 5 years from treatment start.

DETAILED DESCRIPTION:
The trial combines two (Gemcitabine and Atezolizumab). Gemcitabine, alone or in combination regimens is a standard of care for several solid tumors, such as advanced or metastatic NSCLC. It is also used in an off-label setting for pre-treated MPM or naïve MPM in combination with platin-chemotherapy.

Atezolizumab is approved in the United States, European Union and in Switzerland for the treatment of NSCLC, urothelial carcinoma, small cell lung cancer (SCLC), triple-negative breast cancer (TNBC) and hepatocellular carcinoma (HCC) patients.

A significant number of patients with malignant pleural mesothelioma (MPM) and non-small cell lung cancer (NSCLC) are not cured with available treatments and will eventually relapse. After relapse treatment options are limited. Preclinical in vitro studies have demonstrated a synergism of immunotherapy with PD(L)1-targeting monoclonal antibodies and gemcitabine administered in different tumors models and ongoing clinical studies showed encouraging results. This may represent a safe and effective therapy for patients who relapsed or did not respond to standard therapies.

Patients will be treated with gemcitabine (1000 mg/m2 i.v. on day 1 and day 8 of each cycle, (every 3 weeks) and with atezolizumab (1200 mg i.v. on day 1 of each cycle, (every 3 weeks). The trial treatments will be continued for max. 2 years or until discontinuation criteria are met. The follow-up phase will last up to 5 years from treatment start.

The main objective of this trial is to determine the efficacy of chemotherapy (gemcitabine) combined with immunotherapy (atezolizumab) in patients with progressive NSCLC and MPM.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH/GCP regulations before registration and prior to any trial specific procedures including screening procedures.
* For Cohort 1 (NSCLC): Patients with histologically- or cytologically- confirmed squamous or non-squamous metastatic NSCLC stage IIIB-IV (based on TNM classification). Patients must have experienced disease recurrence or progression during or after one or more prior immunotherapy or chemo-immunotherapy regimen for metastatic disease.
* For Cohort 2 (MPM): Patients with histologically confirmed inoperable malignant pleural mesothelioma (MPM; with or without metastasis; all histological subtypes are eligible). Participants must have experienced disease recurrence or progression during or after one or more prior systemic therapy regimen for advanced or metastatic disease.
* Patients with treated and stable CNS metastases are eligible, if:

  * Previous CNS-directed therapy has been completed at least 4 weeks prior to treatment start
  * No evidence of progression after completion of CNS-directed therapy as ascertained by clinical examination and brain imaging (MRI or CT).
* Patients with known HIV-infection are eligible, if:

  * CD4+ T-cell counts are ≥ 350 cells/ųl
  * No history of AIDS-defining opportunistic infection within past 12 months
  * Patient agrees to concomitant antiretroviral therapy (ART) if not currently on ART, or is on ART for ˃ 4 weeks and has a HIV viral load ˂ 400 copies/ml.
* Patients with a previously treated malignancy are eligible if this is clinically stable and does not require concurrent tumor-directed treatment.

Exception: patients suffering from prostate cancer under hormonal ablation therapy (hormone sensitive disease) are eligible.

* Patients with measurable disease according to RECIST 1.1 or mRECIST 1.1.
* Availability of samples for translational research prior to treatment start. For the tumor samples either archival or freshly prepared biopsy samples (cytology is not allowed) are acceptable. Acceptable samples include core needle biopsies for deep tumor tissue (three cores; or in case only two cores can be obtained, there has to be tissue available in order to send 10 unstained slides considered by the local pathologist to be representative of the tumor) or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions.
* Age ≥ 18 years.
* ECOG performance status 0-2.
* Adequate bone marrow function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 90 g/L or ≥ 5.6 mmol/L.
* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), AST and ALT ≤ 2.5 x ULN, or ≤ 5 x ULN for patients with hepatic metastasis.
* Adequate renal function: estimated glomerular filtration rate (eGFR) ≥ 40 ml/min/1.73 m2 (according to the Chronic Kidney Disease Epidemiology Collaboration) abbreviated formula CKD-EPI formula).
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must use highly effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and until 5 months after the last dose of investigational drug. A negative serum or urine pregnancy test before starting of trial treatment is required for all women of childbearing potential.
* Men agree not to donate sperm or to father a child during trial treatment and until 5 months after the last dose of investigational drug (www.swissmedicinfo.ch).
* Patients consent to the mandatory translational research projects providing the required samples.

Exclusion criteria

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Symptomatic brain metastases indicative of active disease (defined as new and/or progressive brain metastases at the time of treatment start [38]) or leptomeningeal disease.
* Prior treatment with gemcitabine in combination with atezolizumab.
* NSCLC patients who progressed within the first 8 weeks from start of first line treatment.
* NSCLC patients with activating EGFR or ALK mutations.
* Known unstable or unresolved surgical or chemotherapy-related toxicity that would compromise trial treatment' duration.
* Concomitant or recent anti-cancer treatment (within 14 days prior to trial treatment start) with any other experimental drug (enrollment in another clinical trial).
* Concomitant use of other anti-cancer drugs or radiotherapy (except for local pain control).
* Cardiac disease NYHA 2 or greater.
* Major surgery within 1 month prior to trial treatment start.
* Known history of any uncontrolled active systemic infection requiring intravenous (i.v.) antimicrobial treatment.
* Known history of tuberculosis, of primary immunodeficiency, of allogeneic tissue/solid organ transplant, of receipt of live attenuated vaccine within 28 days prior to treatment start.
* History of interstitial lung disease (ILD) or severe pneumonitis (other than chronic obstructive pulmonary disease -COPD- exacerbation) that have required oral or i.v. steroids, or uncontrolled pleural effusion.
* Concomitant use of systemic corticosteroids as premedication for chemotherapy.
* Concomitant or prior use of systemic immunosuppressive medication (such as interferon, methotrexate) within 28 days prior to trial treatment start, with the exceptions local (i.e. intranasal, inhaled and topical) corticosteroids.
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information or to the Investigator' Brochure.
* Known or suspected hypersensitivity to trial drug(s) or to any component of the trial drug(s).
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Primary endpoint for cohort 1: Objective response rate (ORR) according to RECIST 1.1 | At the date of tumor assessment according to RECIST 1.1, assessed up to 2 years after registration
  ORR according to RECIST 1.1 is defined as the proportion of patients, whose best overall response is either complete response (CR) or partial response (PR) achieved during trial treatment until disease progression according to RECIST 1.1.
  Patients with CR or PR as best observed response during trial treatment will be considered as success; otherwise as failures for this endpoint.
  Patients without any tumor assessment or with non-evaluable response (NE) during trial treatment will be considered as failures for this endpoint.
Primary endpoint for cohort 2: ORR according to mRECIST | At the date of tumor assessment according to mRECIST, assessed up to 2 years after registration
  ORR according to mRECIST is defined as the proportion of patients, whose best overall response is either complete response (CR) or partial response (PR) achieved during trial treatment until disease progression according to mRECIST.
  Patients with CR or PR as best observed response during trial treatment will be considered as success; otherwise as failures for this endpoint.
  Patients without any tumor assessment or with non-evaluable response (NE) during trial treatment will be considered as failures for this endpoint.

SECONDARY OUTCOMES:
For cohort 1 (NSCLC): Duration of response (DoR) according to RECIST 1.1 | From the time from the first documentation of CR or PR (whichever occurs first) until disease progression according to RECIST 1.1 or death due to any cause, assessed up to 5 years after registration
  DoR according to RECIST 1.1 is defined as the time from the first documentation of CR or PR (whichever occurs first) until disease progression according to RECIST 1.1 or death due to any cause.
  Patients not experiencing an event at the time of analysis and those starting a subsequent treatment without an event will be censored at the date of their last available tumor assessment before starting subsequent treatment, if any.
  This endpoint will be calculated for the subgroup of patients achieving CR or PR.
For cohort 1 (NSCLC): Progression-free survival (PFS) according to RECIST 1.1 | From the date of first dose of atezolizumab/gemcitabine until the date of progressive disease according to RECIST 1.1 or death due to any cause, whichever occurs first, assessed up to 5 years after the first registration
  PFS according to RECIST 1.1 is measured as the time from the first dose of atezolizumab/gemcitabine until disease progression according to RECIST 1.1 or death due to any cause.
  Patients not experiencing an event at the time of analysis and those receiving a subsequent treatment without an event will be censored at the date of their last available tumor assessment before starting subsequent treatment, if any.
For cohort 1 (NSCLC): Disease control rate (DCR) at 18 weeks according to RECIST 1.1 | At the date of tumor assessment according to RECIST 1.1, assessed up to 2 years after registration
  DCR at 18 weeks according to RECIST 1.1 is defined as the proportion of patients, whose best overall response is either CR, PR or stable disease maintained for at least 18 weeks (SD≥18weeks) during trial treatment until disease progression according to RECIST 1.1.
  Patients with CR, PR, SD≥18weeks as best observed response during the trial treatment until disease progression according to RECIST 1.1 will be considered as success; otherwise as failures for this endpoint.
  Patients without any tumor assessment or with non-evaluable response (NE) during trial treatment will be considered as failures for this endpoint.
For cohort 2 (MPM): ORR according to mRECIST 1.1 | At the date of tumor assessment according to mRECIST 1.1, assessed up to 2 years after registration
  ORR according to mRECIST 1.1 is defined as the proportion of patients whose best overall response is either CR or PR achieved during trial treatment until disease progression according to mRECIST 1.1.
  Patients with CR or PR as best observed response will be considered as success; otherwise as failures for this endpoint.
  Patients without any tumor assessment or with non-evaluable response (NE) during trial treatment will be considered as failures for this endpoint.
For cohort 2 (MPM): DoR according to mRECIST 1.1 | From the time from the first documentation of CR or PR (whichever occurs first) until disease progression according to mRECIST 1.1 or death due to any cause, assessed up to 5 years after registration
  DoR according to mRECIST 1.1 is defined as the time from the first documentation of CR or PR (whichever occurs first) until disease progression according to mRECIST 1.1 or death due to any cause, whichever occurs first.
  Patients not experiencing an event at the time of analysis and those starting a subsequent treatment without an event will be censored at the date of their last available tumor assessment before starting subsequent treatment, if any.
  This endpoint will be calculated for the subgroup of patients achieving CR or PR.
For cohort 2 (MPM): PFS according to mRECIST 1.1 | From the date of first dose of atezolizumab/gemcitabine until the date of progressive disease according to mRECIST 1.1 or death due to any cause, whichever occurs first, assessed up to 5 years after registration
  PFS is defined as the time from the first dose of atezolizumab/gemcitabine until disease progression according to mRECIST 1.1 or death due to any cause.
  Patients not experiencing an event at the time of analysis and those receiving a subsequent treatment without an event will be censored at the date of their last available tumor assessment before starting subsequent treatment, if any.
For cohort 2 (MPM): DCR at 18 weeks according to mRECIST 1.1 | At the date of tumor assessment according to mRECIST 1.1, assessed up to 2 years after registration
  DCR at 18 weeks according to mRECIST 1.1 is defined as the proportion of patients whose confirmed best overall response is either CR, PR or stable disease maintained for at least 18 weeks (SD≥18weeks) during trial treatment until disease progression according to mRECIST 1.1.
  Patients with CR, PR, SD18weeks as best observed response will be considered as success; otherwise as failures for this endpoint.
  Patients without any tumor assessment or with non-evaluable response (NE) during trial treatment will be considered as failures for this endpoint.
For cohort 1 and cohort 2: Objective response rate according to iRECIST (iORR) | At the date of tumor assessment according to iRECIST, assessed up to 2 years after registration
  iORR is defined as the proportion of patients whose best overall response is either (CR/iCR) or (PR/iPR) according to RECIST 1.1, modified RECIST 1.1 or iRECIST achieved during trial treatment until disease progression according to iRECIST.
  Patients with CR/iCR or PR/iPR as best observed response during trial treatment until disease progression according to iRECIST will be considered as a success; otherwise as failures for this endpoint.
  Patients without any tumor assessment or with non-evaluable response (NE) during trial treatment will be considered as failures for this endpoint.
For cohort 1 and cohort 2: DoR according to iRECIST (iDoR) | From the time of documentation of CR or PR (whichever occurs first) until disease progression according to iRECIST or death due to any cause, assessed up to 5 years after registration
  iDoR is defined as the time from the first documentation of CR/iCR or PR/iPR (whichever occurs first) according to RECIST 1.1, modified RECIST 1.1 or iRECIST achieved during trial treatment until disease progression according to iRECIST or death due to any cause.
  Patients not experiencing an event at the time of analysis and those starting a subsequent treatment without an event will be censored at the date of their last available tumor assessment before starting subsequent treatment, if any.
  This endpoint will be calculated for the subgroup of patients achieving CR/iCR or PR/iPR.
For cohort 1 and cohort 2: PFS according to iRECIST (iPFS) | From the date of first dose of treatment until the date of progressive disease according to iRECIST or death due to any cause, whichever occurs first, assessed up to 5 years after registration
  iPFS is defined as the time from the first dose of atezolizumab/gemcitabine until disease progression according to iRECIST or death due to any cause.
  Patients not experiencing an event at the time of analysis and those receiving a subsequent treatment without an event will be censored at the date of their last available tumor assessment before starting subsequent treatment, if any.
For cohort 1 and cohort 2: Overall Survival (OS) | From the date of from the first dose of atezolizumab/gemcitabine until the date of death from any cause, assessed up to 5 years after registration
  OS is defined as the time from the first dose of atezolizumab/gemcitabine until death due to any cause. Patients alive or lost to follow-up will be censored at the last date where they were known to be alive.
For cohort 1 and cohort 2: Adverse events (AEs) will be assessed according to CTCAE v5.0. | Up to 5 years after registration
  AEs will be assessed according to CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Curioni Fontecedro, MD, Study Chair — University of Zurich
Locations (12):
- Switzerland (12):
  - HFR Fribourg, Fribourg, Villars-sur-Glâne
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - St. Claraspital, Basel
  - Inselspital, Bern
  - Kantonsspital Graubuenden, Chur
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - UniversitätsSpital Zürich, Zurich
  - Klinik Hirslanden Onkozentrum Zürich, Zurich